CLINICAL TRIAL: NCT03552731
Title: Evaluation of Depression and Anxiety in Chemotherapy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Richmond University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RUMCPSY-ONC
Record Dates: First submitted 2018-05-07; First posted 2018-06-12 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Oncology Problem
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subsequent: Patients who have been receiving chemotherapy more than once. A intervention survey will be administered.
  Interventions: Behavioral: Surveys
- First Time: Patients who have been receiving chemotherapy first time. A intervention survey will be administered.
  Interventions: Behavioral: Surveys

INTERVENTIONS:
Behavioral: Surveys — GAD 7 Survey and PHQ 9 Interventional survey will be administered in both groups.

SUMMARY:
This study will examine the existence and severity of depression and anxiety in patients undergoing chemotherapy at RUMC. Patients currently undergoing initial chemotherapy cycle will be compared to patients undergoing a subsequent chemotherapy cycle. Data will then be collected using standardized depression and anxiety scales to assess if these comorbidities exist and to what severity level. Data already collected for depression and anxiety in patients with chronic, but not cancer, illness will be used as a control.

The participants will be screened for signs of psychological distress using three self administered questionnaires: the Generalized Anxiety Disorder 7 item Scale (GAD7) and Patient Health Questionnaire (PHQ9). Demographic information about the participants, including medical and psychiatric history, will also be gathered from their medical records.

DETAILED DESCRIPTION:
The purpose of the study is to see how common Anxiety, Depression and distress are in people who are undergoing treatment for cancer. We want to understand how common these issues are in order to better screen for, and treat people suffering from them. Past studies have shown that people with anxiety or depression and cancer have worse outcomes, and a study evaluating how common these issues are has not been done. Patients presenting for chemotherapy will be identified and approached for participation by members of the research team. The purpose and design of the study will be explained. After informed consent is obtained, the surveys will be administered by the study team. Completing surveys will take 20 minuets. Relevant demographic information will be collected from the patients EMR. Recruitment will extend over one year period. Those determined to be suffering from anxiety or depression will be given the option of psychiatric follow up or intervention.

ELIGIBILITY:
Inclusion Criteria:1)Patients (greater than equal to) 18 years of age 2)Patients with a confirmed diagnosis of a solid tumor or hematologic cancer 3)Patients who are able to understand the informed consent and read the selfadministered metrics. 4)Patients undergoing chemotherapy.

-

Exclusion Criteria:

* Patients unable to give informed consent.
* Patients with a previous diagnosis of anxiety or depression prior to chemotherapy

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults receiving chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Screener (GAD-7) | Two years
  Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder (GAD). GAD-7 consists total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively. Using the threshold score of 10, the GAD-7 has a sensitivity of 89% and a specificity of 82% for generalized anxiety disorder.

SECONDARY OUTCOMES:
Patient Heath Questionnaire-9 (PHQ-9) | Two years
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: The PHQ-9 incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool.Depression Severity: 0- none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against an independent structured mental health professional (MHP) interview. PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression.

OTHER OUTCOMES:
Demographic Information | Two years
  To gather demographic information with a Demographic Survey

CONTACTS AND LOCATIONS:
Overall Officials: Jakey Patwari, MD, Study Director — Richmond University Medical Center
Locations (1):
- Richmond University Medical Center, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: No